CLINICAL TRIAL: NCT03318380
Title: Contrast-Enhanced Ultrasound Evaluation of Focal Liver Lesions in Patients With Cirrhosis or Other Risk Factors for Developing HCC
Brief Title: Contrast-Enhanced Ultrasound Imaging in Diagnosing Liver Cancer in Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); GE Healthcare (Industry); Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17F.310; JT 10635 (Other: JeffTrial Number); 1R01CA215520-01A1 (NIH)
Record Dates: First submitted 2017-10-12; First posted 2017-10-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic Contrast-Enhanced Ultrasound Imaging (CEUS) (Experimental): Patients receive sulfur hexafluoride IV and undergo CEUS imaging over 10 minutes.
  Interventions: Procedure: Dynamic Contrast-Enhanced Ultrasound Imaging

INTERVENTIONS:
Procedure: Dynamic Contrast-Enhanced Ultrasound Imaging — Undergo CEUS

SUMMARY:
This clinical trial studies how well contrast-enhanced ultrasound imaging works in diagnosing liver cancer in patients with cirrhosis. Diagnostic procedures, such as contrast-enhanced ultrasound imaging, may help find and diagnose liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the sensitivity, specificity, positive and negative predictive values of contrast-enhanced ultrasound (CEUS) for diagnosis of hepatocellular carcinoma (HCC) in patients at risk for HCC in a multicenter setting.

SECONDARY OBJECTIVES:

I. To validate CEUS Liver Imaging Reporting and Data System (LI-RADS) and determine the prevalence of HCC in each CEUS LI-RADS category.

II. To evaluate inter-reader reliability of CEUS for HCC diagnosis. III. To evaluate covariates that might limit diagnostic performance of CEUS for HCC diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Capable of making informed decisions regarding his/her treatment
* Have known cirrhosis or other risk factors for HCC, based on American Association for the Study of Liver Diseases (AASLD) and European Association for the Study of the Liver (EASL) guidelines (applicable in each site jurisdictions)
* Patients with untreated focal liver observations on liver ultrasound or multiphase contrast-enhanced CT or MRI performed as part of clinical standard of care within 4 weeks before patient enrollment.

OR

• Patients with untreated focal liver observations scheduled for follow-up multiphase contrast-enhanced CT or MRI, biopsy or surgical excision as part of clinical standard of care. CEUS should be performed within 4 weeks before or after follow-up imaging or within 4 weeks before biopsy or surgical excision.

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients with focal liver observations less than 5 mm or greater than 5 cm in size
* Patients with contraindications to CEUS
* Patients with contraindications to both CT and MRI
* Patients who are medically unstable, terminally ill, or whose clinical course is unpredictable
* Liver nodule previously treated with trans-arterial or thermal ablation
* Patients who have received an investigational drug in the 30 days before CEUS, or will receive one within 72 hour after their CEUS exam

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity of contrast-enhanced ultrasound evaluation (CEUS) for diagnosis of Hepatocellular cancer using a 95% confidence interval 95% confidence interval for HCC diagnosis using CEUS LR-5 classification | Up to 12 months
  A value of 67% for sensitivity is expected based on recent meta-analysis studies of CEUS for focal liver mass characterization.
Specificity of contrast-enhanced ultrasound evaluation (CEUS) for diagnosis of Hepatocellular cancer using a 95% confidence interval | Up to 12 months
  A value of 91% for specificity is expected based on recent meta-analysis studies of CEUS for focal liver mass characterization.
Positive Predictive Value of contrast-enhanced ultrasound evaluation (CEUS) for diagnosis of Hepatocellular cancer using a 95% confidence interval | Up to 12 months
  A value of 93% for Positive Predicative Value is expected based on recent meta-analysis studies of CEUS for focal liver mass characterization.
Negative Predictive Value of contrast-enhanced ultrasound evaluation (CEUS) for diagnosis of Hepatocellular cancer using a 95% confidence interval | Up to 12 months
  A value of 60% for Negative predictive value is expected based on recent meta-analysis studies of CEUS for focal liver mass characterization.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Lyshchik, MD, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (11):
- United States (6):
  - University of California San Diego, San Diego, California
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
- University of Calgary, Calgary, Canada
- University of Paris, Paris, France
- University of Bologna, Bologna, Italy
- University of Bern, Bern, Switzerland
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kono Y, Piscaglia F, Wilson SR, Medellin A, Rodgers SK, Planz V, Kamaya A, Fetzer DT, Berzigotti A, Sidhu PS, Wessner CE, Bradigan K, Kuon Yeng Escalante CM, Siu Xiao T, Eisenbrey JR, Forsberg F, Lyshchik A; CEUS LI-RADS Trial Group. Clinical impact of CEUS on non-characterizable observations and observations with intermediate probability of malignancy on CT/MRI in patients at risk for HCC. Abdom Radiol (NY). 2024 Aug;49(8):2639-2649. doi: 10.1007/s00261-024-04305-9. Epub 2024 Jun 11. PMID 38860996
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/